CLINICAL TRIAL: NCT04944017
Title: Ketamine for the Treatment of Depression in Parkinson's Disease (KET-PD)
Brief Title: Ketamine for the Treatment of Depression in Parkinson's Disease
Acronym: KET-PD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Fox (Michael J.) Foundation for Parkinson's Research (Unknown)
Responsible Party: Principal Investigator, Sophie Holmes, Assistant Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2000030394; DO NOT RELEASE (Other: CB)
Record Dates: First submitted 2021-06-22; First posted 2021-06-29 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Parkinson's Disease; Depression
Keywords: Ketamine Treatment
MeSH Terms: conditions — Parkinson Disease; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ketamine Infusion (Experimental): Participants will receive 6 infusions of ketamine (0.5 mg/kg IV, up to 60 mg total) , administered over 40 minutes while on continuous cardiac monitoring and oximetry
  Interventions: Drug: Ketamine Infusion
- Saline Infusion (Placebo Comparator): Participants will receive 6 infusions of placebo (saline IV), administered over 40 minutes while on continuous cardiac monitoring and oximetry
  Interventions: Other: Placebo - Saline Infusion

INTERVENTIONS:
Drug: Ketamine Infusion — Participants will receive 6 infusions of ketamine (0.5 mg/kg IV, up to 60 mg total) , administered over 40 minutes while on continuous cardiac monitoring and oximetry
  Arms: Ketamine Infusion
Other: Placebo - Saline Infusion — Participants will receive 6 infusions of saline administered over 40 minutes while on continuous cardiac monitoring and oximetry
  Arms: Saline Infusion

SUMMARY:
The main purpose of this study is to examine the efficacy and safety of a repeated dosing ketamine infusion paradigm compared to placebo in individuals with PD.

A subset of participants in each arm will undergo baseline and post-treatment PET and fMRI scans, to examine whether changes in synaptic density and reorganization of functional networks underlie ketamine's putative antidepressant effects in PD.

DETAILED DESCRIPTION:
This study will assess the efficacy of ketamine for the treatment of depression in Parkinson's disease (PD), in a parallel, double-blind, placebo controlled randomized clinical trial (RCT). Imaging will be used to examine the mechanistic effects of ketamine treatment. Specifically, the investigators will use positron emission tomography (PET) to measure synaptic density and functional magnetic resonance imaging (fMRI) to measure functional connectivity. The investigators hypothesize that a course of ketamine treatment will result in a significant reduction in depression severity compared to placebo. Mechanistically, ketamine will result in a reorganization of functional networks and an increase in synaptic density.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ages 40-80 years, inclusive
2. Clinical diagnosis of Parkinson's disease, stage 1, 2 or 3 as determined by the Hoehn and Yahr Scale
3. Meet criteria for major depressive disorder (MDD) as determined by the Mini-International Neuropsychiatric Interview (MINI), and at least 15 on the MADRS, which has shown maximum discrimination between depressed and non-depressed PD patients.
4. For women of reproductive potential, use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation, as well as a negative pregnancy test at screening.
5. Abstinence from drugs of abuse, other than alcohol, cannabis, nicotine and caffeine for the duration of the study.
6. Stated willingness to comply with all study procedures and availability for the duration of the study.
7. Provision of signed and dated informed consent form.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Presence of Dementia and a Montreal Cognitive Assessment (MoCA) score of less than 18.
2. A primary psychiatric disorder (as determined by the MINI) except for MDD
3. Active suicidal ideation with intent
4. History of substance dependence in the last 2 years
5. Current substance use disorder, except tobacco use disorder
6. Prior clinical psychiatric treatment with ketamine or prior recreational use of ketamine
7. A history of or current significant medical (e.g. cardiovascular, renal), or neurological (e.g. cerebrovascular, seizure, traumatic brain injury) illness other than PD that is unstable and significantly increase their risk and/or might affect the study objectives, as determined by study physicians
8. Uncontrolled hypertension, defined as average blood pressure greater than or equal to 140 mmHg or an average diastolic blood pressure greater than or equal to 90 mmHg among those patients who have hypertension.
9. Orthostatic hypotension (OH) that presents with symptoms sustained longer than a few minutes (e.g., light-headedness, blurred vision, dizziness, weakness, fatigue) or with syncope. OH is defined by a decrease in systolic blood pressure of 20 mm Hg or a decrease in diastolic blood pressure of 10 mm Hg within 3 minutes of standing compared with blood pressure from the sitting position.
10. Inability to provide written informed consent according to the Yale Human Investigation Committee (HIC) guidelines.
11. Any condition or finding that in the judgement of the PI significantly increases risk or significantly reduces the likelihood of benefit from participation in the study.

    For participation in the PET/fMRI only:
12. Prior radiation exposure for research purposes within such that participation in this study would place them over FDA limits for annual radiation exposure (5 rem per yr)
13. Contraindications to MRI scanning.
14. Presence of a bleeding disorder as determined by the PT/INR (Prothrombin time and international normalized ratio) test

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-11-23 (Actual); Primary Completion 2025-09-24 (Actual); Study Completion 2025-09-24 (Actual)

PRIMARY OUTCOMES:
Change in Depression Severity | Baseline, Week 1, Week 2, and Week 3
  The primary outcome of depression severity post-treatment will be compared between groups using a linear mixed model with group (ketamine, placebo) included as a between-subjects factor and time (baseline, weeks 1, 2, 3) included as a within-subjects factor. The scale used to measure depression severity is called The Montgomery-Åsberg Depression Rating Scale (MADRS). The MADRS is a ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in patients with mood disorders. The overall score ranges from 0 to 60, higher MADRS score indicates more severe depression.

SECONDARY OUTCOMES:
Change in Blood pressure: systolic | Baseline and up to 19 days after last administration of study intervention
  Changes in systolic and diastolic blood pressure determined as clinically significant by the Investigator
Change in Blood pressure: diastolic | Baseline and up to 19 days after last administration of study intervention
  Changes in systolic and diastolic blood pressure determined as clinically significant by the Investigator
Change in Heart rate | Baseline and up to 19 days after last administration of study intervention
  Changes in heart rate determined as clinically significant by the Investigator
Change in Respiration | Baseline and up to 19 days after last administration of study intervention
  Changes in respiration determined as clinically significant by the Investigator
Change in O2 saturation | Baseline and up to 19 days after last administration of study intervention
  Changes in O2 saturation determined as clinically significant by the Investigator
Change in ECG | Baseline and up to 19 days after last administration of study intervention
  Changes in ECG indicating a cardiac event such as an arrhythmia or ischemia determined as clinically significant by the Investigator
Change in CBC with differential | Baseline and up to 19 days after last administration of study intervention
  Changes in CBD with differential determined as clinically significant by the Investigator
Change in complete metabolic panel | Baseline and up to 19 days after last administration of study intervention
  Changes in complete metabolic panel determined as clinically significant by the Investigator
Change in TFTs | Baseline and up to 19 days after last administration of study intervention
  Changes in TFTs determined as clinically significant by the Investigator
Change in routine urinalysis | Baseline and up to 19 days after last administration of study intervention
  Changes in routine urinalysis determined as clinically significant by the Investigator
Adverse events | Baseline and up to 32 days after last administration of study intervention
  Assessed by CTCAE v5.0 and the abbreviated version of the SAFTEE-GI and -SI to assess all body systems
Change in synaptic density | Baseline, Week 3
  The change in synaptic (SV2A) density (measured using [11C]UCB-J PET) between baseline and post-intervention scans will be measured across regions of interest
Change in network function | Baseline, Week 3
  The change in network function will be measured by comparing fMRI functional connectivity between baseline and post-intervention scans

CONTACTS AND LOCATIONS:
Overall Officials: Sophie E. Holmes, PhD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States